CLINICAL TRIAL: NCT05945407
Title: Establishment of a Network Platform for Fertility-sparing in Patients With Endometrial Cancer and Study on Fertility-sparing Therapy for Patients With Stage IA Endometrial Cancer.
Brief Title: Fertility-sparing Therapy for Patients With Stage IA Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Peking Union Medical College Hospital (Other); Third Military Medical University (Other); Tianjin Medical University General Hospital (Other); Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Shengjing Hospital (Other); Beijing Chao Yang Hospital (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Chief physician, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017ECFerSp
Record Dates: First submitted 2023-03-26; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Neoplasms; Endometrial Neoplasm Malignant; Endometrial Neoplasm Malignant Stage I; Carcinoma, Endometrioid; Fertility Preservation
Keywords: Fertility-sparing; Fertility-preserving; Endometrial Carcinoma; Endometrial Cancer; Indication Extension
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma, Endometrioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myometrial invasion group (Experimental): Pelvic enhanced magnetic resonance imaging or transvaginal color Doppler ultrasound suggests that the tumor invades less than one half of the myometrium.
  Interventions: Combination Product: Indication-extended Fertility-sparing Therapy
- No myometrial invasion group (Other): Pelvic enhanced magnetic resonance imaging or transvaginal color Doppler ultrasound suggests that the tumor is limited to the endometrium.
  Interventions: Combination Product: Indication-extended Fertility-sparing Therapy

INTERVENTIONS:
Combination Product: Indication-extended Fertility-sparing Therapy — Patients will receive medroxyprogesterone acetate ("FARLUTAL") 250-500mg/d or megestrol acetate ("YiLiZhi") 160-320mg/d orally. If there is no response after 6 months of treatment, change the regimen to levonorgestrel intrauterine system ("Mirena") and gonadotropin-releasing hormone agonist ("Leuprorelin", "Goserelin" or "Triptorelin") 3.75mg/28d injection subcutaneously. After complete remission, the same regimen will be used for consolidation treatment for another 1-3 months. Subsequently, if the patient has no intention of pregnancy, render maintenance treatment ("Mirena", "Progesterone", "Dydrogesterone", or combined oral contraceptive). Otherwise, the patient will be encouraged to conceive either by an expectation for 3-6 months, or by assisted reproductive technology. Indications for stopping fertility-sparing therapy: 1) disease progression; 2) no response after 9 months of treatment; 3) repeated recurrence; 4) no longer require sparing fertility; 5) serious adverse reactions.

SUMMARY:
The goal of this clinical trial is to explore the feasibility and outcome of fertility-sparing therapy in Stage IA G1-G2 Endometrial Cancer with less than 1/2 myometrial invasion. Researchers will render participants indication-extended fertility-sparing therapy. Researchers will compare the myometrial invasion group with the no myometrial invasion group to see if it is possible to propose an extension indication of fertility-sparing therapy for endometrial cancer.

DETAILED DESCRIPTION:
The study population is patients with Stage IA endometrial adenocarcinoma with no myometrial invasion or less than 1/2 myometrial invasion. The sample size is 57 cases (Myometrial invasion group : No myometrial invasion group = 1 : 2). Follow up every 3-6 months until the end of the fifth year of treatment. The primary outcome measure is the complete remission rate after 9 months of treatment. Secondary outcome measures include complete remission rate (6 months/12 months after initial treatment), complete remission time, recurrence rate (1 year/2 years after complete remission), recurrence time, pregnancy rate (1 year after complete remission), pregnancy outcome, blood molecular biomarkers, pathological markers, adverse reactions, etc.

ELIGIBILITY:
Inclusion Criteria:

* Stage IA (FIGO 2009) ;
* Pathological diagnosis: endometrial adenocarcinoma G1-G2;
* MRI or ultrasound: tumor limited to endometrium or invading less than 1/2 of myometrium；
* 18 years old ≤ Age ≤ 45 years old;
* With a strong desire for fertility preservation；
* Sign the informed consent.

Exclusion Criteria:

* Complicated with any other malignancy；
* Contraindications to conservative treatment；
* Contraindications to progestin use;
* Contraindications to pregnancy, or judged by the researcher to be unfit for pregnancy or delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Based on biological sex.
Enrollment: 57 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 9 months after initial treatment
  No endometrioid carcinoma or any proliferative lesion is found by pathology; imaging examination shows no evidence of a tumor.

SECONDARY OUTCOMES:
complete remission rate | 6 months after initial treatment
  No endometrioid carcinoma or any proliferative lesion is found by pathology; imaging examination shows no evidence of a tumor.
complete remission rate | 12 months after initial treatment
  No endometrioid carcinoma or any proliferative lesion is found by pathology; imaging examination shows no evidence of a tumor.
complete remission time | 12 months after initial treatment
  Time required to achieve complete remission.
recurrence rate | 1 year after complete remission
  After complete remission, there is evidence of recurrence in pathology, and the imaging examination shows that the lesion recurs.
recurrence rate | 2 years after complete remission
  After complete remission, there is evidence of recurrence in pathology, and the imaging examination shows that the lesion recurs.
recurrence time | 2 years after complete remission
  Time of recurrence after complete remission.
pregnancy rate | 1 year after complete remission
  A pregnancy test shows pregnancy after complete remission.
pregnancy time | 1 year after complete remission
  Time of pregnancy.
live birth rate | 1 year after pregnancy
  The live birth rate is defined as the ratio of live births to pregnancies.
CA125 | every 3-6 months until 5 years after initial treatment
  Used as a tumor marker for disease monitoring.
HOMA-IR | every 3-6 months until 5 years after initial treatment
  Homeostasis model assessment of insulin resistance is used as an indicator to evaluate the level of insulin resistance.
pathological markers | every 3-6 months until 5 years after initial treatment
  Immunohistochemical analysis is used to assess the expression of Ki-67, ER/PR, p53, PTEN, and mismatch repair proteins (MLH1, PMS2, MSH2, and MSH6).
adverse reactions | every 3-6 months until 5 years after initial treatment
  Harmful reactions unrelated to the purpose of treatment occur during normal prevention, diagnosis, and treatment of diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Jianliu Wang, Professor, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hosoital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No